CLINICAL TRIAL: NCT06520046
Title: Motor Control Prevention Strategies for Ankle Sprains in Basketball Players
Brief Title: Motor Control Prevention Strategies in Basketball Players
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Rocío Llamas-Ramos, Associate Professor, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MOTORCONTROL2024
Record Dates: First submitted 2024-07-09; First posted 2024-07-25 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-07

CONDITIONS: Ankle Sprains; Motor Disorders
MeSH Terms: conditions — Ankle Injuries; Motor Disorders | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Motor control group (Experimental): Basketball players aged between 10-18 years old who play regularly in one of the basketball sports clubs in the city of Salamanca.
  The study will be carried out in 20 sessions. As for the proprioception and balance work, a simple proposal of exercises will be made, increasing the difficulty from the fifth session onwards. From the 10th session onwards, unstable surfaces will be introduced as long as our athletes are capable of achieving the task of less complexity. If it is not possible to progress in intensity, the same level will be maintained.
  Interventions: Other: Experimental Group
- Control (Active Comparator): Basketball players aged between 10-18 years old who play regularly in one of the basketball sports clubs in the city of Salamanca.
  These participants shall carry out their usual treatment
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Experimental Group — Propioceptive exercises
  Arms: Motor control group
Other: Control Group — Usual exercises
  Arms: Control

SUMMARY:
Ankle sprains have always been considered as isolated injury entities, in which the passive ankle stabilisation system suffered an elongation due to trauma. Today, this concept of an isolated injury has evolved into a more holistic concept, interrelated with various components from different sources.

ELIGIBILITY:
Inclusion Criteria:

* Basketball players aged between 10-18 years old who play regularly in one of the basketball clubs in the city of Salamanca.

Exclusion Criteria:

* previous injuries
* fractures
* use of orthoses and technical aids

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Range of motion | At the beginning and at 9 months
  Measurements of the articular range of the ankle joint
Musculature Strength | At the beginning and at 9 months
  Measurement of the strength of the musculature of the back of the leg by means of isokinetic tests
Presence of Myofascial trigger points | At the beginning and at 9 months
  Diagnostic criteria established by Travell and Simons, the presence or absence of active or latent myofascial trigger points will be assessed.
Speed of contraction of the musculature | At the beginning and at 9 months
  By means of the isokinetic tests and the aforementioned exploratory curves, the speed of contraction of the musculature of the back of the leg and foot will be evaluated

IPD SHARING:
Plan to Share IPD: Undecided